CLINICAL TRIAL: NCT07079605
Title: Cardiac Manifestations of Sepsis and Its Association With Disease Outcome: A Prospective Cohort Study
Brief Title: Sepsis and Myocarditis
Status: Recruiting | Type: Observational
Sponsor: Jimma University (Other)
Collaborators: Ethiopian Society of Cardiac Professionals (Unknown)
Responsible Party: Principal Investigator, Kedir Negesso Tukeni, MD, Internist and cardiologist, PhD fellow in Medical Research, Cardiovascular Science, Jimma University
Other Study IDs: JUIH/IRB/278/25
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Sepsis-related Myocarditis
Keywords: Sepsis; myocarditis; mortality; survival analysis; low in-come countries; Ethiopia
MeSH Terms: conditions — Sepsis; Myocarditis | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: This is a group of patients with the diagnosis of sepsis of any focus but without any signs/symptoms suggestive of cardiac involvement.
  Interventions: Other: Standard treatment for sepsis of any focus
- Group B: This is a cohort of patients with the diagnosis of sepsis of any foci and with the evidences of cardiac involvement defined as one or a combination of the following:
  * Clinical symptoms include chest pain, dyspnea, or arrhythmias.
  * Abnormal biomarkers, including troponins or BNP levels.
  * Evidence of cardiac dysfunction on ECG or echocardiography.
  Both groups will be followed prospectively for 9 to 1 year to evaluate their outcomes.
  Interventions: Other: Treatment for the sepsis with standard management of cardiac failure

INTERVENTIONS:
Other: Standard treatment for sepsis of any focus — This group of patients will be treated for the sepsis of any focus as per standard.
  Groups: Group A
Other: Treatment for the sepsis with standard management of cardiac failure — This group of patients will be treated for the sepsis and management of cardiac failure with additional supportive care cocktails based on the specific indication.
  Groups: Group B

SUMMARY:
This prospective cohort study aims to investigate the cardiac manifestations of sepsis and their influence on disease outcomes among adult patients at Jimma University Medical Center, Ethiopia, from May 2025 to May 2026. The research will include adults aged 18 and older with sepsis, categorizing them based on the presence or absence of cardiac involvement, which will be assessed through clinical symptoms, biomarkers, ECG, and echocardiographic findings. The study will evaluate the persistence of cardiac abnormalities, functional capacity, and survival over one year, utilizing structured data collection and advanced statistical methods, including survival analysis and regression techniques, to identify predictors of adverse outcomes.

DETAILED DESCRIPTION:
Background: Sepsis is a major cause of morbidity and mortality worldwide, frequently associated with multi-organ dysfunction, including the heart. Cardiac manifestations of sepsis, such as myocardial dysfunction and arrhythmias, significantly impact outcomes, yet their long-term implications remain inadequately studied, particularly in resource-limited settings like Ethiopia.

Objective: The objective of this study is to evaluate the cardiac manifestations of sepsis and their association with disease outcomes among adult patients with sepsis at Jimma University Medical Centre of Ethiopia.

Methodology: This prospective cohort study will be conducted at JUMC over one-year period, starting from May 2025 to May 2026. The study will be done on adult patients with no prior history of cardiac problems (aged ≥18 years) diagnosed with sepsis (including bacterial meningitis), and then grouped based on the presence (Group A) or absence (Group B) of sepsis-associated cardiac manifestations. Cardiac involvement will be defined using clinical symptoms, biomarkers (troponin, BNP), or abnormal ECG and echocardiographic findings. Outcomes, including persistence of cardiac abnormalities, functional capacity and survival, will be assessed and compared among both groups after one year of follow-up. Data will be gathered using a structured checklist and analysed using updated version software. The Kaplan-Meier curve and the log-rank test will be used to describe the survival function. Independent predictors of poor outcome will be identified by Cox regression analysis, and the model assumption will be checked by Schoenfeld and Cox-Snell residuals. The 95% confidence interval of the hazard ratio with a corresponding p-value of 0.05 will be used to declare statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged 18 years and above diagnosed with sepsis admitted to Jimma University Medical Center during the study periods that are willing to participate and continue follow-up of their disease condition for at least one year.

Exclusion Criteria:

* Patients with any kind of pre-existing established cardiac disease prior to their sepsis diagnosis and those who are not willing to participate or not willing to have follow-up of their disease condition for at least one year.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include all adult septic patients admitted to JUMC during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Composite outcomes of survival status and persistence or resolution of cardiac abnormalities. | at first, third and sixth- months post discharge
  Outcomes will be assessed at the first, third, and sixth months post-discharge, with evaluations focusing on the following parameters:
  * Persistence or resolution of cardiac abnormalities
  * Survival status (alive or deceased)
  * Functional capacity and quality of life using standardized tools (KCCS).

SECONDARY OUTCOMES:
Composite outcomes of persistence or resolution of cardiac abnormalities, Survival status (alive or deceased) and functional capacity and quality of life using standardized tools (KCCS). | at sixth- months post discharge
  Outcomes will be assessed at six months post-discharge, with evaluations focusing on the following parameters:
  * Persistence or resolution of cardiac abnormalities
  * Survival status (alive or deceased)
  * Functional capacity and quality of life using standardized tools (KCCS).

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Alexander Haas, MD, Pediatician, Cardiologist, Study Chair — Ludwig Maximillians University of Munich, Germany
Locations (1):
- Jimma University Hospital, Jimma, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
The team is yet to decide whether to share IPD or not.

REFERENCES:
- [Result] Rudiger A, Singer M. Mechanisms of sepsis-induced cardiac dysfunction. Crit Care Med. 2007 Jun;35(6):1599-608. doi: 10.1097/01.CCM.0000266683.64081.02. PMID 17452940
- [Result] Merx MW, Weber C. Sepsis and the heart. Circulation. 2007 Aug 14;116(7):793-802. doi: 10.1161/CIRCULATIONAHA.106.678359. PMID 17698745
- [Result] Song J, Fang X, Zhou K, Bao H, Li L. Sepsis-induced cardiac dysfunction and pathogenetic mechanisms (Review). Mol Med Rep. 2023 Dec;28(6):227. doi: 10.3892/mmr.2023.13114. Epub 2023 Oct 20. PMID 37859613
- [Result] Habimana R, Choi I, Cho HJ, Kim D, Lee K, Jeong I. Sepsis-induced cardiac dysfunction: a review of pathophysiology. Acute Crit Care. 2020 May;35(2):57-66. doi: 10.4266/acc.2020.00248. Epub 2020 May 31. PMID 32506871
- [Result] Jentzer JC, Lawler PR, Van Houten HK, Yao X, Kashani KB, Dunlay SM. Cardiovascular Events Among Survivors of Sepsis Hospitalization: A Retrospective Cohort Analysis. J Am Heart Assoc. 2023 Feb 7;12(3):e027813. doi: 10.1161/JAHA.122.027813. Epub 2023 Feb 1. PMID 36722388
- [Result] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. No abstract available. PMID 24171518
- [Result] Kwizera A, Urayeneza O, Mujyarugamba P, Baelani I, Meier J, Mer M, Musa N, Kissoon N, Patterson AJ, Farmer JC, Dunser MW. Epidemiology and Outcome of Sepsis in Adults and Children in a Rural, Sub-Sahara African Setting. Crit Care Explor. 2021 Dec 16;3(12):e0592. doi: 10.1097/CCE.0000000000000592. eCollection 2021 Dec. PMID 34939034
- [Result] Mulatu HA, Bayisa T, Worku Y, Lazarus JJ, Woldeyes E, Bacha D, Taye B, Nigussie M, Gebeyehu H, Kebede A. Prevalence and outcome of sepsis and septic shock in intensive care units in Addis Ababa, Ethiopia: A prospective observational study. Afr J Emerg Med. 2021 Mar;11(1):188-195. doi: 10.1016/j.afjem.2020.10.001. Epub 2020 Nov 5. PMID 33680740